CLINICAL TRIAL: NCT00163579
Title: The Impact of the Prophylactic or Therapeutic Application of Bryophyllum on Preterm Delivery - a Prospective Study
Brief Title: The Impact of Bryophyllum on Preterm Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BS-2004-UFK-1; 2004 DR 5192 swissmedic (Other: Swissmedic)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Preterm Delivery; Preterm Contractions; Cervical Shortening
Keywords: premature birth; cerclage; tocolysis; drug therapy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bryophyllum (Experimental)
  Interventions: Drug: Bryophyllum
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bryophyllum
  Arms: Bryophyllum
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is whether Bryophyllum is more effective and has less side effects than traditional labor inhibitors in preventing preterm delivery.

DETAILED DESCRIPTION:
Preterm delivery (delivery before 37 +0 weeks of gestation) is still the leading cause of perinatal mortality and morbidity in the western countries. Due to this fact it is only possible to achieve the mortality rate of 5‰, aspired by WHO, by an effective decrease of the current preterm delivery rate.

An exact ascertainment of the etiology of preterm delivery is hardly possible, because multiple, partly overlapping or multifactorial etiologies exist. Various pathologies (e.g. of the placenta, fetus uterus or endocrine dysfunctions) may lead to preterm deliveries or preterm contractions.

Traditional diagnostic tools for preterm contractions/preterm deliveries has consisted of clinical examinations (digital palpation of the cervix) and the recording of the contractions by the tocogram. Both methods have a low sensitivity and predictive values. Furthermore the clinical examination has a high interobserver variability of 29%.

With the introduction of transvaginal sonographic measurements, the sensitivity for preterm deliveries could substantially be elevated.

Despite intensive efforts in the field of preventive care, screening and therapeutic interventions (e.g. the use of tocolytics), the incidence of preterm deliveries has remained stable for over two decades.

For inhibiting labor, beta-mimetics has been utilised for over 20 years. Beta mimetics are currently able to prevent preterm labor in average for approximately 48 hours. Other medicaments with tocolytic properties include calcium antagonists, prostaglandin inhibitors and currently, antagonists of the oxytocic receptor.

However, conventional labor inhibitors show considerable side effects, such as cardiovascular effects (e.g.tachycardia) or tremor in case of beta mimetics.

Due to the stagnant long-term results of the conventional labor inhibitors, we are looking for alternative medicaments, especially with a lower side effect profile.

The phytopharmacon Bryophyllum, which is produced from the leaves of Bryophyllum pinnatum, is available as a 5% aqueous tincture, 33% dilution or 50% trituration.

Bryophyllum has been used since 1970 for tocolysis, either orally or intravenously. However, because of its predominant use in anthroposophical clinics, clinical trials for its evaluation has been rarely performed. Currently, in vitro studies endorsed the inhibition of myometrial contractibility. In contrast to conventional labor inhibitors, side effects has been only occasionally observed in case of Bryophyllum (e.g. skin irritation).

To evaluate the tocolytic effects of orally applicated Bryophyllum versus Placebo in case of patients with preterm contractions, twin pregnancies and patients with a risk for preterm delivery, due to previous preterm contractions/preterm deliveries.

Bryophyllum or Placebo will be given prophylactic or, parallel with conventional labor inhibitors in case of preterm contractions.

ELIGIBILITY:
Inclusion Criteria:

All multiple pregnancies Singleton pregnancies with preterm contractions/cervix < 25mm, or singleton pregnancies with burdened maternal anamnesis (e.g. prior preterm delivery preterm contractions cerclage).

Exclusion Criteria:

* Fetal malformations
* Chromosomal anomalies
* Intrauterine growth restriction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Extension of pregnancy

SECONDARY OUTCOMES:
Rate of preterm deliveries, rate of side effects, days of hospitalisation, rate of lung maturation.

CONTACTS AND LOCATIONS:
Overall Officials: Irène Hoesli, Prof. Dr. MD, Principal Investigator — Women's University Hospital, Basel, Switzerland
Locations (1):
- Obstetrical Unit, Women's University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Plangger N, Rist L, Zimmermann R, von Mandach U. Intravenous tocolysis with Bryophyllum pinnatum is better tolerated than beta-agonist application. Eur J Obstet Gynecol Reprod Biol. 2006 Feb 1;124(2):168-72. doi: 10.1016/j.ejogrb.2005.05.013. Epub 2005 Jul 26. PMID 16051414
- [Background] Gwehenberger B, Rist L, Huch R, von Mandach U. Effect of Bryophyllum pinnatum versus fenoterol on uterine contractility. Eur J Obstet Gynecol Reprod Biol. 2004 Apr 15;113(2):164-71. doi: 10.1016/S0301-2115(03)00370-1. PMID 15063954
- [Background] Vilaghy I. [Decreasing the rate of premature delivery with phytotherapy--results from general practice]. Ther Umsch. 2002 Dec;59(12):696-701. doi: 10.1024/0040-5930.59.12.696. German. PMID 12584959